CLINICAL TRIAL: NCT04463745
Title: Organ Dysfunction Associated With Intraabdominal Pressures in Liver Transplantation
Brief Title: Organ Dysfunction Associated With Intra Abdominal Pressures in Liver Transplantation
Acronym: OIL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS - Liver Transplant-3
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-09

CONDITIONS: Liver Diseases; Intra-Abdominal Hypertension; Cirrhosis, Liver; Organ Dysfunction Syndrome
Keywords: organ dysfunction; intra-abdominal pressure; liver transplantation; liver cirrhosis
MeSH Terms: conditions — Liver Diseases; Intra-Abdominal Hypertension; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver Transplant Recipients: adult patients undergoing liver transplantation

SUMMARY:
Patients with end stage liver disease have varying degrees of intra-abdominal hypertension (IAH) due to the presence of ascites. The perioperative events may either relieve or aggravate the intra-abdominal pressures. Intra-abdominal hypertension has damaging effect on various organ systems. There is an increase in intracranial pressures and a decrease in cerebral perfusion pressures associated with IAH . In the heart, there is an increase of right atrial pressures, increase in systemic vascular resistance and decrease in cardiac output . Pulmonary complications include increase in the peak, mean and plateau airway pressures, with decreased compliance . Renal dysfunction is an early effect of raised intra-abdominal pressure, resulting from decreased renal blood flow, shunting of blood to the medulla, mechanical compression of the kidneys and increased pressures in the renal veins . We would study the intra-abdominal pressures in liver transplant recipients and record hemodynamic, respiratory, cardiac and renal function prospectively. Follow up data for 6 days for neurological, respiratory, cardiac and renal complications will be collected, along with hospital stay, ICU stay and mortality. The association between intra-abdominal pressures and these outcomes will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing liver transplantation
* 18 to 65 years

Exclusion Criteria:

* pregnant patients
* primary diagnosis of Acute liver failure and acute on chronic liver failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing liver transplantation for various indications , including chronic liver disease due to alcohol, NASH , viral hepatitis among others.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
28 day mortality | 28 days
  mortality of any cause in the fist 28 days after transplantation
duration of icu stay | 28 days
  time period spent in the intensive care unit

SECONDARY OUTCOMES:
Acute kidney injury in 1st week | 7 days
  incidence of acute kidney injury in 1 week of transplantation
Respiratory complications | 7 days
  includes duration of ventilation, incidence of vap
major neurological complications | 7 days
  any major neurological event

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ponnappan, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India